CLINICAL TRIAL: NCT04690218
Title: Evaluation of Sleep Quality, Nutrition, Anxiety and Depression in Mastalgia
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Alirıza Erdoğan, Principal Investigator, Nigde Omer Halisdemir University
Other Study IDs: 2020/86
Record Dates: First submitted 2020-12-26; First posted 2020-12-30 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Mastodynia
Keywords: mastodynia; anxiety; depression; sleep quality
MeSH Terms: conditions — Mastodynia; Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mastalgia: "Mastalgia" group will consist of women with confirmed mastalgia. The patients will be asked to fulfill the forms of Hospital Anxiety and Depression Scale and Pittsburgh Sleep Quality Index. Additionally patients will be asked to inform the frequency and amount of consumption of certain nutritional elements by a questionnaire.
  Interventions: Diagnostic Test: Hospital anxiety and depression scale; Diagnostic Test: Pittsburgh Sleep Quality Index; Behavioral: Nutritional Status Questionnaire
- Controls: "Controls" group will consist of women attending to general surgery clinic for reasons other than mastalgia. The patients will be asked to fulfill the forms of Hospital Anxiety and Depression Scale and Pittsburgh Sleep Quality Index. Additionally patients will be asked to inform the frequency and amount of consumption of certain nutritional elements by a questionnaire.
  Interventions: Diagnostic Test: Hospital anxiety and depression scale; Diagnostic Test: Pittsburgh Sleep Quality Index; Behavioral: Nutritional Status Questionnaire

INTERVENTIONS:
Diagnostic Test: Hospital anxiety and depression scale — Self assessment scale suitable for hospital community as well as public community. Applying the scale does not require any psychopathologic training.
Diagnostic Test: Pittsburgh Sleep Quality Index — Self assessment scale for public community. Applying the scale does not require any specially trained personnel.
Behavioral: Nutritional Status Questionnaire — It consists of 26 items, questioning the frequency and amount of certain nutritional elements (ones known to worsen and benefit mastalgia) consumed by the individual.

SUMMARY:
The aim of this study is to investigate the sleep quality, anxiety and depression levels in women with mastalgia using internationally validated scales. Additionally the investigators aim to question the amount and frequency of consumption of nutritional elements which are known to aggravate mastalgia. Finally by combining and analyzing the information gathered, the investigators intend to set light to the etiopathologic and clinic aspects of mastalgia.

DETAILED DESCRIPTION:
Mastalgia is encountered in 70% of premenopausal women and is one of the most frequent reasons for attending general surgery clinics. In most of the cases no physical cause is demonstrated and the etiopathogenesis is still not yet determined. In 1949 Patey, for the first time, proposed that mastalgia might be a psychologically based problem. In the following years, research was focused in this issue and some articles were published demonstrating the relationship of anxiety, depression and high stress levels with mastalgia. The efforts for finding out the etiopathologic mechanism and defining the risk factors revealed that smoking and consumption of tea, coffee and carbonated beverages in particular worsen mastalgia whereas essential fatty acids (especially gamma linoleic acid) provides a symptomatic relief. Additionally it is known that sleep irregularities cause serious deterioration in daily life quality as well as can exaggerate some medical, neurologic and/or psychiatric conditions. More than half of the population experience sleep irregularities from time to time and chronic sleep disturbances effect 20% of adult population in western countries. Therefore sleep irregularities might have contributing effects in the etiopathogenesis and/or symptomatology of therapy resistant conditions like mastalgia.

ELIGIBILITY:
Inclusion Criteria:

* Having mastalgia as a presenting symptom (mastalgia group)
* Presence of mastalgia confirmed by a general surgeon (mastalgia group)
* Absence of mastalgia (control group)

Exclusion Criteria:

* Previously diagnosed breast carcinoma (both groups)
* Previously exposed to thoracic radiotherapy (both groups)
* Previous breast or thoracic surgery for any reason (both groups)
* Presence of Tietze syndrome (both groups)
* Use of nutritional supplements (both groups)
* Presence of any self-perceived pain (control group)
* Presence of psychogenic based conditions and psychosomatic illnesses (control group)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Mastalgia group (women with mastalgia) and controls (women without mastalgia)
Study Population: This case-controlled study will consist of 2 groups; Mastalgia group (women with confirmed mastalgia) and controls (women without mastalgia).
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Score | 9 months
  Hospital Anxiety and Depression Score is four point likert type scale. It consists of 14 questions. Questions 1, 3, 5, 7, 9, 11 and 13 address anxiety whereas questions 2, 4, 6, 8, 10, 12 and 14 address depression. Achievable minimum score of the scale is 0 and the maximum score is 42. The cut-off score for depression is 7 and for anxiety is 10. Scores higher than 7 indicate high anxiety levels and scores higher than 10 indicate the presence of depression.
Pittsburgh Sleep Quality Index | 9 months
  Pittsburgh Sleep Quality Index consists of 7 component. The possible scoring range of the scale is 0-21. The high scores indicates bad sleep quality. The cutt-off value is 5.
The amount of nutritional elements consumed which worsen mastalgia | 9 months
  Calculated as the number stated by the individual (times consumed per day/week/month)

SECONDARY OUTCOMES:
The amount of other nutritional elements consumed | 9 months
  Calculated as the number stated by the individual (times consumed per day/week/month)

CONTACTS AND LOCATIONS:
Locations (1):
- Niğde Ömer Halisdemir University Training and Research Hospital, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kanat BH, Atmaca M, Girgin M, Ilhan YS, Bozdag A, Ozkan Z, Yazar FM, Emir S. Effects of Mastalgia in Young Women on Quality of Life, Depression, and Anxiety Levels. Indian J Surg. 2016 Apr;78(2):96-9. doi: 10.1007/s12262-015-1325-5. Epub 2015 Aug 28. PMID 27303116
- [Background] PATEY DH. Two common non-malignant conditions of the breast; the clinical features of cystic disease and the pain syndrome. Br Med J. 1949 Jan 15;1(4593):96-9. doi: 10.1136/bmj.1.4593.96. No abstract available. PMID 18122751
- [Background] Preece PE, Mansel RE, Hughes LE. Mastalgia: psychoneurosis or organic disease? Br Med J. 1978 Jan 7;1(6104):29-30. doi: 10.1136/bmj.1.6104.29. PMID 620138
- [Background] Johnson KM, Bradley KA, Bush K, Gardella C, Dobie DJ, Laya MB. Frequency of mastalgia among women veterans. Association with psychiatric conditions and unexplained pain syndromes. J Gen Intern Med. 2006 Mar;21 Suppl 3(Suppl 3):S70-5. doi: 10.1111/j.1525-1497.2006.00378.x. PMID 16637950
- [Background] Colegrave S, Holcombe C, Salmon P. Psychological characteristics of women presenting with breast pain. J Psychosom Res. 2001 Jun;50(6):303-7. doi: 10.1016/s0022-3999(01)00196-9. PMID 11438111
- [Background] Ader DN, South-Paul J, Adera T, Deuster PA. Cyclical mastalgia: prevalence and associated health and behavioral factors. J Psychosom Obstet Gynaecol. 2001 Jun;22(2):71-6. doi: 10.3109/01674820109049956. PMID 11446156
- [Background] Idiz C, Cakir C, Ulusoy AI, Idiz UO. The Role of Nutrition in Women with Benign Cyclic Mastalgia: A Case-Control Study. Eur J Breast Health. 2018 Jul 1;14(3):156-159. doi: 10.5152/ejbh.2018.3827. eCollection 2018 Jul. PMID 30123881
- [Background] Soldatos CR, Paparrigopoulos TJ. Sleep physiology and pathology: pertinence to psychiatry. Int Rev Psychiatry. 2005 Aug;17(4):213-28. doi: 10.1080/09540260500104565. PMID 16194793
- [Background] Barthlen GM, Stacy C. Dyssomnias, parasomnias, and sleep disorders associated with medical and psychiatric diseases. Mt Sinai J Med. 1994 Mar;61(2):139-59. PMID 8022426
- [Background] Mollayeva T, Thurairajah P, Burton K, Mollayeva S, Shapiro CM, Colantonio A. The Pittsburgh sleep quality index as a screening tool for sleep dysfunction in clinical and non-clinical samples: A systematic review and meta-analysis. Sleep Med Rev. 2016 Feb;25:52-73. doi: 10.1016/j.smrv.2015.01.009. Epub 2015 Feb 17. PMID 26163057
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771